CLINICAL TRIAL: NCT05930275
Title: A Multi-country, Prospective, Post-marketing Study of UPadacitinib Evaluating Speed of Onset and Durability of Effectiveness for Patients With Moderate to Severe Crohn's Disease for 3 Years in Real-world Clinical Practice (UPlift)
Brief Title: Study to Assess Speed of Onset and Durability of Effectiveness of Upadacitinib in Adult Participants With Moderate to Severe Crohn's Disease (CD) in Real World Clinical Practice.
Acronym: UPlift
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-899
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; CD; Upadacitinib
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label.

SUMMARY:
Crohn's disease (CD) is an incurable chronic inflammatory disorder of the gastrointestinal tract. This study will assess how safe and effective upadacitinib is in treating moderately to severely active CD in real world. Speed of onset and durability of effectiveness will be assessed.

Upadacitinib is a drug approved for the treatment of CD. All study participants will receive upadacitinib as prescribed by their study doctor in accordance with approved local label. Approximately 1200 participants will be enrolled in approximately 230 sites across the world.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 3 years.

There is expected to be no additional burden for participants in this trial. Study visits may be conducted on-site or virtually as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of moderate-to-severe crohn's disease (CD).
* Participants initiating upadacitinib at the clinician's discretion as part of their routine clinical care; the decision to administer upadacitinib must be made prior to and independent of recruitment into the study.
* Participants prescribed upadacitinib in accordance with the approved local label.
* Able to understand and communicate with the investigator and comply with the requirements of the study.
* Willing to continue with study documentation after cessation of upadacitinib.
* Willing and able to participate in the collection of PRO data via a cloud-based application on their personal or provided mobile phone or website app.

Exclusion Criteria:

* Any contraindication to upadacitinib.
* Previously exposure to upadacitinib in a clinical trial.
* Currently participating in interventional research (not including non-interventional study, post-marketing observational study (PMOS) , or registry participation).
* Initiation of upadacitinib prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with Crohn's disease (CD)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Time to Achieve First Clinical Response (CR) per Patient-Reported Outcome 2 (PRO2) (Daily CR-PRO) | Up to Week 12
  Daily CR-PRO is a composite endpoint defined as the first day with at least 30% decrease in daily very soft or liquid stool frequency (SF) and/or >= 30% decrease in daily abdominal pain (AP) score and both not worse than baseline and a prospective 7-day average daily CR-PRO starting on the first day of daily CR-PRO; prospective 7-day average daily CR-PRO is defined as >= 30% decrease in average daily very soft or liquid SF and/or >= 30% decrease in average daily AP score and both not worse than baseline.
Percentage of Participants Achieving Clinical Remission per Harvey Bradshaw Index (HBI) Among those with Clinical Response-Harvey Bradshaw Index (CR-HBI) at End of Induction Therapy | At Week 52
  Clinical Remission is defined as HBI <= 4. Clinical Response is defined as HBI reduction >= 3 points from baseline. The HBI is a simplified version of the Crohn's Disease Activity Index(CDAI). The HBI consists of 5 items encompassing patient reported (well-being, symptoms) and objective (presence of abdominal mass or complications) variables. The total HBI score is the sum of the values for each of the five items. Higher HBI scores indicate greater disease activity. Scores < 5 indicate clinical remission, 5 - 7 indicate mild disease activity, 8 - 16 indicate moderate disease activity, and 16 indicate severe disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (180):
- Australia (7):
  - Blacktown Hospital /ID# 258574, Blacktown, New South Wales
  - Macquarie University Hospital /ID# 268722, Macquarie University, New South Wales
  - Mater Misericordiae Limited /ID# 258535, South Brisbane, Queensland
  - Ibd Sa /Id# 268335, Kurralta Park, South Australia
  - The Queen Elizabeth Hospital /ID# 258536, Woodville South, South Australia
  - Monash Health - Monash Medical Centre /ID# 258538, Clayton, Victoria
  - The Alfred Hospital /ID# 258537, Melbourne, Victoria
- Bulgaria (9):
  - Gastro Med EOOD /ID# 267777, Pazardzhik, Plovdiv
  - ET dr Nikolay Tsonev /ID# 267584, Samokov, Sofia
  - MC Higia HB /ID# 267575, Sofiya, Sofia
  - Umbal Kaspela /ID# 267562, Plovdiv
  - Diagnostic consultative center Focus-5 /ID# 267576, Sofia
  - Diagnostic consultative center Focus-5 /ID# 268600, Sofia
  - AIPSMP dr Mirchev EOOD /ID# 267583, Varna
  - MC Nadejda Femily EOOD /ID# 267585, Varna
  - DCC Mladost M /ID# 267586, Varna
- Canada (15):
  - Foothills Medical Centre /ID# 263475, Calgary, Alberta
  - Dr. J Siffledeen Profess Pract /ID# 262713, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 262347, New Westminster, British Columbia
  - University of Manitoba & Shared Health /ID# 265853, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre - Victoria General /ID# 262764, Halifax, Nova Scotia
  - Barrie GI Associates /ID# 268436, Barrie, Ontario
  - London Health Sciences Center- University Hospital /ID# 262693, London, Ontario
  - West GTA Endoscopy /ID# 262946, Mississauga, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 262060, North Bay, Ontario
  - Toronto Immune and Digestive Health Institute Inc /ID# 262540, North York, Ontario
  - ABP Research Services Corp. /ID# 263111, Oakville, Ontario
  - Toronto Digestive Disease Associates /ID# 262050, Vaughan, Ontario
  - Universite de Montreal - Hopital Maisonneuve-Rosemont /ID# 266264, Montreal, Quebec
  - Disc_Royal Victoria Hospital / McGill University Health Centre /ID# 262692, Montreal, Quebec
  - Diex Recherche Quebec Inc. /ID# 268256, Québec
- China (9):
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 265873, Beijing, Beijing Municipality
  - Chongqing General Hospital /ID# 268384, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun-Yat Sen University /ID# 264189, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 265673, Guangzhou, Guangdong
  - Nanjing Drum Tower Hospital /ID# 266205, Nanjing, Jiangsu
  - Ruijin Hospital /ID# 266869, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University /ID# 265674, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital /ID# 270703, Chengdu, Sichuan
  - Jinhua Central Hospital /ID# 265871, Jinhua, Zhejiang
- Czechia (3):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 268351, Brno, Brno-mesto
  - SurGal Clinic /ID# 268757, Brno, South Moravian
  - Nemocnice Ceske Budejovice /ID# 264492, České Budějovice
- Denmark (2):
  - Herlev Hospital /ID# 262487, Herlev, Capital Region
  - Hvidovre Hospital /ID# 262613, Hvidovre, Capital Region
- Estonia (3):
  - West Tallinn Central Hospital /ID# 270144, Tallinn, Harju
  - East Tallinn Central Hospital - Magdaleena Unit /ID# 266653, Tallinn, Harju
  - Tartu University Hospital /ID# 270148, Tartu, Tartu
- France (27):
  - Chu de Nice-Hopital L'Archet Ii /Id# 261060, Nice, Alpes-Maritimes
  - CHU Clermont-Ferrand /ID# 259294, Clermont, Auvergne-Rhône-Alpes
  - Hopital Edouard Herriot /ID# 266844, Lyon, Auvergne-Rhône-Alpes
  - APHM - Hopital Nord /ID# 259304, Marseille, Bouches-du-Rhone
  - Chu Dijon /Id# 265910, Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Universitaire de Bordeaux /ID# 259298, Pessac, Gironde
  - CHU Toulouse - Hopital Rangueil /ID# 258636, Toulouse, Haute-Garonne
  - Clinique Beau Soleil /ID# 259289, Montpellier, Herault
  - CHU de Montpellier - Hopital Saint Eloi /ID# 269938, Montpellier, Herault
  - Ch Chalons En Champagne /Id# 259344, Châlons-en-Champagne, Marne
  - CHRU Lille - Hopital Claude Huriez /ID# 259302, Lille, Nord
  - Cabinet du docteur Médina Boualit /ID# 259291, Saint-Amand-les-Eaux, Nord
  - AP-HP - Hopital Bicetre /ID# 259118, Le Kremlin-Bicêtre, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 259293, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 259303, St-Priest-en-Jarez, Pays de la Loire Region
  - Centre Hospitalier de la Cote Basque /ID# 259297, Bayonne, Pyrenees-Atlantiques
  - GH Mutualiste Les Portes Du Sud /ID# 259299, Vénissieux, Rhone
  - Hôpital Nord Ouest - Villefranche-sur-Saône /ID# 266999, Villefranche-sur-Saône, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 259121, Amiens, Somme
  - Pole Sante Saint-Jean /ID# 259296, Cagnes-sur-Mer
  - Centre Hospitalier de CHOLET /ID# 259288, Cholet
  - CH DREUX - Hopital Victor Jousselin /ID# 258635, Dreux
  - AP-HP - Hopital Saint-Antoine /ID# 259116, Paris
  - CHRU Pontchaillou /ID# 259347, Rennes
  - CHU de Strasbourg /ID# 259343, Strasbourg
  - Hopital Beaujon /ID# 259287, Clichy, Île-de-France Region
  - Centre Medico Chirurgical Ambroise Pare Hartmann /ID# 259339, Neuilly-sur-Seine, Île-de-France Region
- Germany (18):
  - Medizinisches Versorgungszentrum Dachau /ID# 273294, Dachau, Bavaria
  - Klinikum Lueneburg /ID# 256107, Lüneburg, Lower Saxony
  - Verein für Wissenschaft und Forschung /ID# 265880, Oldenburg, Lower Saxony
  - Dres. Kamp & Partner /ID# 267560, Minden, North Rhine-Westphalia
  - Praxis S. Tetzlaff /ID# 264613, Buedelsdorf, Schleswig-Holstein
  - Praxis fuer Gastroenterologie /ID# 256106, Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Jena /ID# 273284, Jena, Thuringia
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 264097, Berlin
  - Gastro Studien GbR /ID# 264617, Berlin
  - Krankenhaus Waldfriede /ID# 264616, Berlin
  - Dr. Janschek /ID# 273218, Dresden
  - SKH Studien GmbH /ID# 256100, Hamburg
  - Private Practice - Dr. Matthias Eichler /ID# 256105, Hamburg
  - Medizinische Hochschule Hannover /ID# 256109, Hanover
  - GSGH Gastroenterologische Studiengesellschaft Herne GbR /ID# 268434, Herne
  - Gastropraxis Magdeburg /ID# 266789, Magdeburg
  - Praxis Dres Brendel /ID# 256103, Nuremberg
  - Praxis Dr. Kempelmann /ID# 256110, Tostedt
- Greece (10):
  - Evangelismos Hospital /ID# 268132, Athens, Attica
  - General Hospital of Athens G. Gennimatas /ID# 271501, Athens, Attica
  - General Hospital of Athens Ippokratio /ID# 270248, Athens, Attica
  - General Hospital of Athens Laiko /ID# 266262, Athens, Attica
  - University General Hospital of Heraklion /ID# 266260, Heraklion, Crete
  - University General Hospital of Alexandroupoli /ID# 270161, Alexandroupoli, Evros
  - Sotiria Thoracic Diseases Hospital of Athens /ID# 264352, Athens
  - General Hospital of Athens Alexandra /ID# 266261, Athens
  - General State Hospital of Nikaia /ID# 264351, Athens
  - Hippokration General Hospital of Thessaloniki /ID# 264353, Thessaloniki
- Hungary (5):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 258518, Debrecen, Hajdú-Bihar
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 258517, Szombathely, Vas County
  - Semmelweis Egyetem /ID# 258515, Budapest
  - Eszak-Pesti Centrumkorhaz - Honvedkorhaz /ID# 267156, Budapest
  - Szegedi Tudományegyetem /ID# 258514, Szeged
- Ireland (3):
  - Portiuncula University Hospital /ID# 268856, Ballinasloe, Galway
  - St. Vincent's University Hospital /ID# 265638, Dublin
  - Connolly Hospital /ID# 266388, Dublin
- Italy (8):
  - Azienda Ospedaliero Universitaria di Cagliari - P.O. Duilio Casula /ID# 268732, Monserrato, Cagliari
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 269224, San Giovanni Rotondo, Foggia
  - IRCCS Istituto Clinico Humanitas /ID# 268731, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 268426, Milan, Milano
  - Fondazione IRCCS San Gerardo dei Tintori - Ospedale San Gerardo /ID# 269589, Monza, Monza E Brianza
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 268759, Rome, Roma
  - A.O. Ordine Mauriziano di Torino /ID# 269231, Turin, Torino
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 275093, Palermo
- Japan (34):
  - Nagoya University Hospital /ID# 266092, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 266091, Toyoake, Aichi-ken
  - Hirosaki University Hospital /ID# 266065, Hirosaki, Aomori
  - Chiba University Hospital /ID# 266080, Chiba, Chiba
  - Toho University Sakura Medical Center /ID# 266079, Sakura, Chiba
  - Kyushu University Hospital /ID# 266100, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 266071, Fukushima, Fukushima
  - Asahikawa Medical University Hospital /ID# 266062, Asahikawa-shi, Hokkaido
  - Asahikawa Medical University Hospital /ID# 269111, Asahikawa-shi, Hokkaido
  - Sapporo Medical University Hospital /ID# 265042, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 266063, Sapporo, Hokkaido
  - Hyogo Medical University Hospital /ID# 266097, Nishinomiya, Hyōgo
  - University of Tsukuba Hospital /ID# 266075, Tsukuba, Ibaraki
  - Iwate Medical University - Yahaba Campus /ID# 266067, Hizume, Iwate
  - Yokohama City University Medical Center /ID# 266087, Yokohama, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID# 268258, Kyoto, Kyoto
  - Kansai Medical University Hospital /ID# 266095, Hirakata-shi, Osaka
  - Saga University Hospital /ID# 267884, Saga, Saga-ken
  - Saitama Medical Center /ID# 266078, Kawagoe, Saitama
  - Shiga University of Medical Science /ID# 266094, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 266090, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital /ID# 266077, Shimotsuke-shi, Tochigi
  - Tokyo Medical And Dental University Hospital /ID# 266081, Bunkyo-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 266084, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 266086, Mitaka-shi, Tokyo
  - Keio University Hospital /ID# 266085, Shinjuku-ku, Tokyo
  - Fukuoka University Hospital /ID# 266099, Fukuoka
  - Hiroshima University Hospital /ID# 266098, Hiroshima
  - Osaka Police Hospital /ID# 266096, Osaka
  - Sapporo Kosei General Hospital /ID# 266069, Sapporo
  - The Jikei University School of Medicine /ID# 266083, Tokyo
  - Tokyo Yamate Medical Center /ID# 266082, Tokyo
  - Toyama University Hospital /ID# 266089, Toyama
  - Toyama Prefectural Central Hospital /ID# 266088, Toyama
- Netherlands (4):
  - Radboudumc /ID# 264659, Nijmegen, Gelderland
  - Elisabeth TweeSteden Ziekenhuis /ID# 265898, Tilburg, North Brabant
  - OLVG - Locatie Oost /ID# 267099, Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC /ID# 253970, Amsterdam, North Holland
- Romania (11):
  - Fundeni Clinical Institute /ID# 260354, Bucharest, București
  - Fundeni Clinical Institute /ID# 260356, Bucharest, București
  - Fundeni Clinical Institute /ID# 264021, Bucharest, București
  - Spitalul Universitar de Urgență București /ID# 263763, Bucharest, București
  - Spitalul Universitar de Urgență București /ID# 264025, Bucharest, București
  - Spitalul Clinic Judetean de Urgenta Craiova /Id# 264023, Craiova, Dolj
  - Spitalul Clinic Colentina /ID# 260355, Bucharest
  - Gastromond /ID# 263770, Constanța
  - Spitalul Clinic Județean de Urgențe "Sfântul Spiridon" /ID# 264022, Iași
  - Spitalul Clinic Județean de Urgențe "Sfântul Spiridon" /ID# 264024, Iași
  - Cabinet Particular Policlinic Algomed /ID# 260353, Timișoara
- Spain (12):
  - Hospital de Sant Joan Despí Moisès Broggi /ID# 263936, Sant Joan Despí, Barcelona
  - Hospital Jerez De La Frontera /ID# 273598, Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofia /ID# 263461, Córdoba, Cordoba
  - Hospital Universitario de Gran Canaria Doctor Negrín /ID# 263462, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Severo Ochoa /ID# 263933, Leganés, Madrid
  - Hospital Universitario Central de Asturias /ID# 263457, Oviedo, Principality of Asturias
  - Hospital Galdakao-Usansolo /ID# 263458, Galdakao, Vizcaya
  - Hospital Universitari Vall d'Hebron /ID# 263463, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 264206, Granada
  - Hospital Universitario de La Princesa /ID# 263464, Madrid
  - Hospital General Universitario Reina Sofía /ID# 264205, Murcia
  - Hospital Alvaro Cunqueiro /ID# 263460, Pontevedra

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P23-899